CLINICAL TRIAL: NCT03708328
Title: An Open Label, Multicenter, Dose Escalation and Expansion, Phase 1 Study to Evaluate Safety, Pharmacokinetics, and Preliminary Anti-Tumor Activity of RO7121661, a PD-1/TIM-3 Bispecific Antibody, in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: A Dose Escalation and Expansion Study of Lomvastomig, a PD-1/TIM-3 Bispecific Antibody, in Participants With Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP40435; 2018-000982-35 (EudraCT Number)
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors; Metastatic Melanoma; Non-small Cell Lung Cancer (NSCLC); Small Cell Lung Cancer (SCLC); Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Part A: Once Every 2 Weeks (Q2W) (Experimental): Lomvastomig will be administered in treatment cycles once every 2 weeks (Q2W). Dose escalation will be carried out according to a modified continual reassessment method (mCRM) with escalation with overdose control (EWOC) design.
  Interventions: Drug: Lomvastomig
- Expansion Part B1: Metastatic Melanoma Cohort (Experimental): This cohort will comprise participants with checkpoint inhibitor (CPI) experienced, second line and beyond metastatic melanoma. The starting dose of lomvastomig for Expansion will be derived from the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: Lomvastomig
- Expansion Part B2: NSCLC Cohort 1 (Experimental): This cohort will comprise participants with CPI and platinum experienced, second or third line PD-L1 positive non-small cell lung cancer (NSCLC). The starting dose of lomvastomig for Expansion will be derived from the MTD/RDE and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: Lomvastomig
- Expansion Part B3: NSCLC Cohort 2 (Experimental): This cohort will comprise participants with PD-L1 high, cancer immunotherapy (CIT) naïve first line NSCLC. The starting dose of lomvastomig for Expansion will be derived from the MTD/RDE and the best dosing schedule determined during Dose Escalation.
  This cohort was not initiated and no participants were enrolled in it.
  Interventions: Drug: Lomvastomig
- Expansion Part B4: SCLC Cohort (Experimental): This cohort will comprise participants with CPI naïve small cell lung cancer (SCLC) with prior failure of, progression on, or intolerance to, standard therapy. The starting dose of lomvastomig for Expansion will be derived from the MTD/RDE and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: Lomvastomig
- Expansion Part B5: ESCC Cohort (Experimental): This cohort will comprise participants with CPI-naïve esophageal squamous cell carcinoma (ESCC). The starting dose of lomvastomig for Expansion will be derived from the MTD/RDE and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: Lomvastomig

INTERVENTIONS:
Drug: Lomvastomig — Lomvastomig will be administered intravenously (IV) with a flat dose on the schedule described for each study arm.
  Other Names: RO7121661; RG7769

SUMMARY:
This is a first-in-human, open-label, multicenter, Phase I multiple-ascending dose (MAD) study of single agent lomvastomig (RO7121661), an anti PD-1 (programmed death-1) and TIM-3 (T-cell immunoglobulin and mucin domain 3) bispecific antibody, for participants with advanced and/or metastatic solid tumors. The study consists of 2 parts: Dose Escalation (Part A) and Expansion (Parts B1, B2, B3, B4, and B5). The Dose Escalation part will be conducted first to determine the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) based on safety, tolerability, pharmacokinetic, and/or the pharmacodynamic profile of escalating doses of lomvastomig. The Expansion part will enroll tumor-specific cohorts to evaluate anti-tumor activity of the MTD and/or RDE of lomvastomig from Part A (Q2W) and to confirm safety and tolerability in participants with selected tumor types.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Part A: Patient must have histologically or cytologically confirmed advanced and/or metastatic solid tumor malignancies for which standard curative or palliative measures do not exist, are no longer effective, or are not acceptable to the patient
* Eastern Cooperative Oncology Group Performance Status 0-1
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
* Fresh biopsies may be required
* Negative HIV, hepatitis B, or hepatitis C test result
* Women of childbearing potential and male participants must agree to remain abstinent or use contraceptive methods as defined by the protocol

Additional Specific Inclusion Criteria for Participants with Melanoma:

* Histologically confirmed, unresectable stage III or stage IV melanoma
* Previously treated with approved anti-programmed death-ligand 1 (PD-L1)/anti-programmed death-1 (PD-1) agents with or without approved anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) therapy and up to one additional treatment regimen

Additional Specific Inclusion Criteria for Participants with Non-small Cell Lung Cancer (NSCLC) who Previously Received Treatment for Metastatic Disease:

* Histologically confirmed advanced NSCLC
* Previously treated with approved PD-L1/PD-1 inhibitors and platinum-based chemotherapy
* Not more than 2 prior lines of treatment for metastatic disease are allowed prior to enrolling to the study
* Participants must have experienced initial clinical benefit (stable disease or better) from most recent checkpoint inhibitor (CPI) therapy
* Tumor PD-L1 expression as determined by immunohistochemistry assay of archival tumor tissue or tissue obtained at screening

Additional Specific Inclusion Criteria for Participants with Non-small Cell Lung Cancer (NSCLC) who Previously Did Not Receive Treatment for Metastatic Disease:

* Histologically confirmed advanced NSCLC
* Tumor PD-L1 expression as determined by immunohistochemistry assay of archival tumor tissue or tissue obtained at screening

Additional Specific Inclusion Criteria for Participants with Small Cell Lung Cancer (SCLC):

* Histologically confirmed SCLC
* Participants may have had prior chemotherapy, radiation therapy, or declined approved therapies for SCLC

Additional Specific Inclusion Criteria for Participants with Esophageal Squamous Cell Carcinoma (ESCC):

* Participants whose major lesion was histologically confirmed as squamous cell carcinoma or adenosquamous cell carcinoma of the esophagus
* Patients who have previously received not more than 1 prior line of treatment for metastatic disease prior to enrolling to the study

Exclusion Criteria:

General Exclusion Criteria:

* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to any of the components of RO7121661
* Active or untreated central nervous system (CNS) metastases
* An active second malignancy
* Evidence of concomitant diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infection
* Treatment with oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* Active or history of autoimmune disease or immune deficiency
* Prior treatment with adoptive cell therapies, such as CAR-T therapies
* Concurrent therapy with any other investigational drug <28 days or 5 half-lives of the drug, whichever is shorter, prior to the first RO7247669 administration
* Regular immunosuppressive therapy
* Radiotherapy within the last 4 weeks before start of study drug treatment, with the exception of limited palliative radiotherapy
* Prior treatment with a T-cell immunoglobulin and mucin domain-3 (TIM-3) inhibitor

Additional Specific Exclusion Criteria for Participants with NSCLC who Previously Received Treatment for Metastatic Disease:

- Patients with the following mutations, rearrangements, translocations are not eligible: epidermal growth factor receptor (EGFR); anaplastic lymphoma kinase (ALK); ROS proto-oncogene 1 (ROS1), BRAFV600E, and neurotrophic receptor tyrosine kinase (NTRK)

Additional Specific Exclusion Criteria for Participants with NSCLC who Did Not Previously Receive Treatment for Metastatic Disease:

* Prior therapy for metastatic disease
* Adjuvant anti-PD-1 or anti-PD-L1 therapy

Additional Specific Exclusion Criteria for Participants with Small-Cell Lung Cancer (SCLC):

- Prior therapy with any immune CPIs (such as anti-PD-L1/PD-1, CTLA-4)

Additional Specific Exclusion Criteria for Participants with Esophageal Squamous Cell Carcinoma (ESCC):

- Prior therapy with any immunomodulatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (2):
  - Columbia Univ Med Ctr, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Denmark (2):
  - Herlev Hospital, Herlev
  - Rigshospitalet, København Ø
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU Timone, Marseille
  - ICO Rene Gauducheau, Saint-Herblain
- Auckland City Hospital, Auckland, New Zealand
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 134 participants with advanced and/or metastatic solid tumors took part in the study across 17 investigative sites in Spain, France, Republic of Korea, Denmark, United States and New Zealand from 15 October 2018 to 09 July 2024.
Pre-assignment Details: This study was conducted in two parts: Part A (Dose Escalation) and Part B (Tumor-Specific Expansion Cohorts). Part B included the Cohorts B1, B2, B4, and B5, enrolling participants with selected tumor types. Part B3 was not initiated.
Groups:
- Part A: Lomvastomig 70 mg: Participants received 70 milligrams (mg) of lomvastomig, as an intravenous (IV) infusion on Cycle 1 Day 1 and every two weeks (Q2W) thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part A: Lomvastomig 210 mg: Participants received 210 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part A: Lomvastomig 615 mg: Participants received 615 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part A: Lomvastomig 1200 mg: Participants received 1200 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part A: Lomvastomig 1800 mg: Participants received 1800 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part A: Lomvastomig 2100 mg: Participants received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B1: Metastatic Melanoma Expansion Cohort: Participants with checkpoint inhibitor (CPI) experienced second line and beyond metastatic melanoma received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B2: NSCLC Expansion Cohort 1: Participants with CPI and platinum experienced second- or third-line programmed death-ligand 1 (PD-L1) positive non-small cell lung cancer (NSCLC) received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B4: SCLC Expansion Cohort: Participants with CPI-naïve SCLC with prior failure of, progression on, or intolerance to standard therapy received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B5: ESCC Expansion Cohort: Participants with CPI-naïve ESCC received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
Period: Overall Study
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Started | 3 | 5 | 4 | 4 | 4 | 19 | 38 | 26 | 15 | 16
Completed | 0 | 1 | 0 | 1 | 1 | 1 | 7 | 2 | 0 | 2
Not Completed | 3 | 4 | 4 | 3 | 3 | 18 | 31 | 24 | 15 | 14
Not completed — Death | 3 | 3 | 4 | 2 | 2 | 13 | 26 | 18 | 13 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 5
Not completed — Study Closed Locally | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Ended By Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Participant Was Alive, Did Not Return to Hospital | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Part A: Lomvastomig 70 mg: Participants received 70 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Total: Total of all reporting groups
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort | Total
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19 | 38 | 26 | 15 | 16 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.3) | 59.6 (13.9) | 61.0 (2.4) | 53.8 (7.1) | 53.5 (15.8) | 60.9 (8.8) | 61.1 (12.1) | 62.3 (9.7) | 60.3 (9.2) | 61.1 (10.6) | 60.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 2 | 9 | 17 | 11 | 1 | 4 | 49
  Male | 2 | 4 | 3 | 2 | 2 | 10 | 21 | 15 | 14 | 12 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 2 | 5 | 3 | 2 | 4 | 17 | 28 | 20 | 15 | 8 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 0 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 8 | 2 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 5 | 4 | 4 | 4 | 18 | 28 | 14 | 13 | 4 | 97
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 0 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: A DLT was defined as a clinically significant adverse event (AE) or significant laboratory abnormality: 1) occurring during DLT assessment period of 21 days; 2) considered to be related to study treatment RO7121661 by the Investigator; 3) is not attributed to disease progression or another clearly identifiable cause. Following AEs were considered DLTs: Hematological toxicities (Grade 4 neutropenia lasting >5 days, Grade ≥3 febrile neutropenia, Grade 4 thrombocytopenia lasting > 48 hours, Grade 3 thrombocytopenia associated with bleeding episodes, Grade 4 anemia, Grade ≥3 anemia with hemolysis); Non-hematological toxicity Grade ≥3 (Any Grade 3 immune-mediated AE, Grade 3 hyperbilirubinemia lasting for >48 hours/Grade 4 hyperbilirubinemia; Grade ≥3 aspartate aminotransferase (AST) or alanine aminotransferase (ALT) elevations with hyperbilirubinemia of Grade ≥2, Grade 4 AST or ALT elevations, Grade ≥3 nausea, vomiting, or diarrhea, Grade ≥3 non-hematological laboratory abnormality.
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 7 (Cycle length= 14 days)
Population: The DLT-evaluable population included all participants in Part A who received at least two doses of study medication and either experienced a DLT within the DLT period or cleared the DLT period without a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19
Participants | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With at Least One AE by Highest Severity, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: AE=any untoward medical occurrence in a participant administered a pharmaceutical product & which does not necessarily have a causal relationship with treatment & can therefore be any unfavorable & unintended sign (including abnormal laboratory values/abnormal clinical test results), symptoms/disease temporally associated with the use of pharmaceutical product, whether or not considered related to pharmaceutical product. Severity of AEs was graded as: Grade 1=Mild, asymptomatic/mild symptoms, clinical/diagnostic observations only, or intervention not indicated; Grade 2=Moderate, minimal, local/non-invasive intervention indicated, or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe/medically significant but not immediately life-threatening, hospitalization/prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4= Life-threatening consequences, urgent intervention indicated; Grade 5=Death related to AE.
Time Frame: From signing of informed consent form up to 60 days after last treatment administration (up to 41.7 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19
Participants
  AEs (Any grade) | 3 | 5 | 4 | 4 | 3 | 18
  Grade 1 AE | 0 | 3 | 1 | 0 | 0 | 2
  Grade 2 AE | 2 | 1 | 2 | 2 | 1 | 9
  Grade 3 AE | 1 | 1 | 1 | 1 | 2 | 7
  Grade 4 AE | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Part B: Objective Response Rate (ORR) as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as the percentage of participants with an objective tumor response of complete response (CR) or partial response (PR) as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: Cycle 1 Day 1 then every 8 weeks for the first year; every 12 weeks thereafter until disease progression or treatment discontinuation (whichever occurs last), initiation of a new line of therapy or death (Up to 43.3 months) (Cycle length= 14 days)
Population: Efficacy population included all participants in the safety population who received at least one dose of study drug and who had at least one baseline and one on-study tumor assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Part B4: SCLC Expansion Cohort: Participants with CPI-naïve small cell lung cancer (SCLC) with prior failure of, progression on, or intolerance to standard therapy received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B5: ESCC Expansion Cohort: Participants with CPI-naïve esophageal squamous cell carcinoma (ESCC) received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 38 | 25 | 15 | 15
percentage of participants | 7.9 (2.19) [2.19 to 19.16] | 0 (0.00) [0.00 to 11.29] | 0 (0.00) [0.00 to 18.10] | 20.0 (5.68) [5.68 to 43.98]

4. Primary Outcome: Part B: Disease Control Rate (DCR) as Determined by Investigator Using RECIST v1.1
Description: DCR was defined as the percentage of participants with an objective tumor response of CR, PR or stable disease (SD) as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression (PD). PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 38 | 25 | 15 | 15
percentage of participants | 36.8 (23.83) [23.83 to 51.47] | 36.0 (20.24) [20.24 to 54.39] | 0 (0.00) [0.00 to 18.10] | 60.0 (35.96) [35.96 to 80.91]

5. Primary Outcome: Part B: Duration of Response (DOR) as Determined by Investigator Using RECIST v1.1
Description: DOR was calculated for participants who had a best confirmed overall response (OR) of CR/PR. DOR was defined as time from first occurrence of a documented OR until the time of documented PD or death (within 30 days from last treatment) from any cause, whichever occurs first as determined by investigator assessment using RECIST v1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Data for participants without PD or death as of the data cut-off date were censored at the time of the last tumor assessment.
Time Frame: From first occurrence of documented OR up to disease progression or death (Up to 43.3 months) (Cycle length = 14 days)
Population: Efficacy population included all participants in the safety population who received at least one dose of study drug and who had at least one baseline and one on-study tumor assessment. Overall number analyzed is the number of participants with OR, i.e., responders.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 0 | 0 | 3
months | 17.7 [3.9 to NA] — The upper limit of the 90% confidence interval (CI) was not estimable due to insufficient number of participants with events. |  |  | 10.6 [3.9 to NA] — The upper limit of the 90% CI was not estimable due to insufficient number of participants with events.

6. Primary Outcome: Part B: Progression Free Survival (PFS) as Determined by Investigator Using RECIST v1.1
Description: PFS was defined as the time from study treatment initiation (Cycle 1 Day 1) to the first occurrence of documented PD, as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Data for participants without PD or death as of the data cut-off date were censored at the time of the last tumor assessment.
Time Frame: From treatment initiation (Cycle 1 Day 1) until disease progression or death (Up to 43.3 months) (Cycle length= 14 days)
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 38 | 25 | 15 | 15
months | 1.8 (1.7) [1.7 to 2.0] | 1.7 (1.6) [1.6 to 1.9] | 1.7 (1.6) [1.6 to 1.8] | 3.6 (1.5) [1.5 to 5.7]

7. Secondary Outcome: Parts A and B: Number of Participants With Treatment Emergent Anti-Drug Antibodies (ADAs)
Description: Participants were considered to be ADA positive if they were ADA negative at baseline but developed an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples was greater than the titer of the baseline sample by a scientifically reasonable margin such as at least 4-fold (treatment-enhanced ADA response).
Time Frame: Baseline and Day 1 of Cycles 1 to 5; Day 1 of Cycle 7, and every 6 cycles thereafter (1 cycle is 14 days); study completion/discontinuation; safety follow-up visits (up to approximately 40.8 months - Part A and 45.4 months - Part B)
Population: Safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. The number of participants analyzed for each group indicates the number of participants with an ADA assay result from at least one post-baseline sample.
Measure: Count of Participants; unit: Participants
Groups:
- Part B1: Metastatic Melanoma Expansion Cohort: Participants with checkpoint inhibitor (CPI) experienced second line and beyond metastatic melanoma received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B2: NSCLC Expansion Cohort 1: Participants with CPI and platinum experienced second- or third-line programmed death-ligand 1 (PD-L1) positive non-small cell lung cancer (NSCLC) received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B4: SCLC Expansion Cohort: Participants with CPI-naïve small cell lung cancer (SCLC) with prior failure of, progression on, or intolerance to standard therapy received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B5: ESCC Expansion Cohort: Participants with CPI-naïve esophageal squamous cell carcinoma (ESCC) received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 3 | 3 | 17 | 37 | 25 | 14 | 16
Participants | 3 | 2 | 0 | 0 | 1 | 3 | 5 | 7 | 1 | 6

8. Secondary Outcome: Part B: Biomarkers: T-cell Proliferation/Activation in Peripheral Blood
Description: Biomarker analyses were performed using peripheral blood samples that were collected from participants in Part B of the study. The blood samples were assessed by flow cytometry for absolute counts of CD3⁺CD8⁺ T cells and proliferating CD3⁺CD8⁺Ki67⁺ T cells.
Time Frame: Days 1, 2, and 8 of Cycles 1 and 5; Day 1 of Cycles 2, 3, and 9 (1 cycle is 14 days); study completion visit (28 days after last dose; up to 43.3 months); safety follow-up (SFU) (90 days after last dose; up to 45.4 months)
Population: The safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Overall number analyzed = participants with data available for analysis. Number analyzed = participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 37 | 26 | 15 | 2
cells per microliter (cells/µL)
  CD3+CD8+: Cycle 1 Day 1: number analyzed (Participants) | 32 | 24 | 15 | 2
  CD3+CD8+: Cycle 1 Day 1 | 350.63 (186.81) | 293.25 (137.62) | 252.60 (224.48) | 256.00 (138.59)
  CD3+CD8+: Cycle 1 Day 2: number analyzed (Participants) | 36 | 25 | 15 | 2
  CD3+CD8+: Cycle 1 Day 2 | 371.61 (219.58) | 317.28 (175.47) | 296.20 (519.44) | 306.50 (111.02)
  CD3+CD8+: Cycle 1 Day 8: number analyzed (Participants) | 32 | 22 | 15 | 1
  CD3+CD8+: Cycle 1 Day 8 | 364.09 (264.35) | 342.59 (223.74) | 292.47 (349.48) | 329.00 (NA) — Since only 1 participant was analyzed, the standard deviation (SD) could not be calculated.
  CD3+CD8+: Cycle 2 Day 1: number analyzed (Participants) | 35 | 23 | 15 | 2
  CD3+CD8+: Cycle 2 Day 1 | 378.54 (250.58) | 298.91 (153.88) | 245.93 (226.21) | 257.00 (66.47)
  CD3+CD8+: Cycle 3 Day 1: number analyzed (Participants) | 32 | 17 | 11 | 1
  CD3+CD8+: Cycle 3 Day 1 | 422.00 (380.62) | 310.47 (171.87) | 193.18 (81.24) | 199.00 (NA) — Since only 1 participant was analyzed, the SD could not be calculated.
  CD3+CD8+: Cycle 5 Day 1: number analyzed (Participants) | 17 | 8 | 4 | 0
  CD3+CD8+: Cycle 5 Day 1 | 403.88 (270.34) | 269.00 (106.32) | 234.00 (72.48) |
  CD3+CD8+: Cycle 5 Day 2: number analyzed (Participants) | 17 | 7 | 4 | 0
  CD3+CD8+: Cycle 5 Day 2 | 445.53 (228.03) | 285.71 (120.35) | 260.50 (59.52) |
  CD3+CD8+: Cycle 5 Day 8: number analyzed (Participants) | 15 | 7 | 3 | 0
  CD3+CD8+: Cycle 5 Day 8 | 516.80 (332.31) | 267.57 (116.42) | 179.00 (68.02) |
  CD3+CD8+: Cycle 9 Day 1: number analyzed (Participants) | 11 | 0 | 1 | 0
  CD3+CD8+: Cycle 9 Day 1 | 503.91 (425.19) |  | 237.00 (NA) — Since only 1 participant was analyzed, the SD could not be calculated. |
  CD3+CD8+: SFU: number analyzed (Participants) | 8 | 2 | 2 | 0
  CD3+CD8+: SFU | 429.38 (302.79) | 453.00 (212.13) | 201.00 (209.30) |
  CD3+CD8+: Study Completion: number analyzed (Participants) | 20 | 12 | 5 | 0
  CD3+CD8+: Study Completion | 296.70 (177.13) | 289.83 (168.98) | 193.80 (136.60) |
  CD3+CD8+Ki67+: Cycle 1 Day 1: number analyzed (Participants) | 31 | 23 | 14 | 2
  CD3+CD8+Ki67+: Cycle 1 Day 1 | 12.45 (8.64) | 11.83 (8.67) | 7.36 (5.51) | 5.50 (2.12)
  CD3+CD8+Ki67+: Cycle 1 Day 2: number analyzed (Participants) | 36 | 23 | 14 | 2
  CD3+CD8+Ki67+: Cycle 1 Day 2 | 13.94 (16.29) | 13.00 (12.76) | 7.71 (7.45) | 8.00 (2.83)
  CD3+CD8+Ki67+: Cycle 1 Day 8: number analyzed (Participants) | 32 | 22 | 14 | 1
  CD3+CD8+Ki67+: Cycle 1 Day 8 | 14.34 (11.67) | 13.64 (12.62) | 11.00 (4.88) | 13.00 (NA) — Since only 1 participant was analyzed, the SD could not be calculated.
  CD3+CD8+Ki67+: Cycle 2 Day 1: number analyzed (Participants) | 33 | 23 | 15 | 2
  CD3+CD8+Ki67+: Cycle 2 Day 1 | 18.12 (22.33) | 17.52 (23.14) | 14.87 (6.62) | 8.50 (0.71)
  CD3+CD8+Ki67+: Cycle 3 Day 1: number analyzed (Participants) | 31 | 17 | 11 | 1
  CD3+CD8+Ki67+: Cycle 3 Day 1 | 16.10 (23.21) | 13.41 (9.21) | 13.45 (8.71) | 8.00 (NA) — Since only 1 participant was analyzed, the SD could not be calculated.
  CD3+CD8+Ki67+: Cycle 5 Day 1: number analyzed (Participants) | 15 | 8 | 3 | 0
  CD3+CD8+Ki67+: Cycle 5 Day 1 | 16.27 (12.27) | 6.88 (2.42) | 9.00 (1.73) |
  CD3+CD8+Ki67+: Cycle 5 Day 2: number analyzed (Participants) | 16 | 6 | 4 | 0
  CD3+CD8+Ki67+: Cycle 5 Day 2 | 19.63 (26.26) | 7.83 (4.17) | 6.75 (2.22) |
  CD3+CD8+Ki67+: Cycle 5 Day 8: number analyzed (Participants) | 15 | 7 | 3 | 0
  CD3+CD8+Ki67+: Cycle 5 Day 8 | 15.33 (9.98) | 7.00 (2.08) | 6.67 (3.79) |
  CD3+CD8+Ki67+: Cycle 9 Day 1: number analyzed (Participants) | 11 | 0 | 1 | 0
  CD3+CD8+Ki67+: Cycle 9 Day 1 | 14.27 (12.58) |  | 6.00 (NA) — Since only 1 participant was analyzed, the SD could not be calculated. |
  CD3+CD8+Ki67+: SFU: number analyzed (Participants) | 8 | 2 | 2 | 0
  CD3+CD8+Ki67+: SFU | 15.63 (12.93) | 22.50 (14.85) | 7.50 (7.78) |
  CD3+CD8+Ki67+: Study Completion: number analyzed (Participants) | 19 | 12 | 5 | 0
  CD3+CD8+Ki67+: Study Completion | 10.58 (7.80) | 9.58 (10.49) | 14.80 (9.31) |

9. Secondary Outcome: Part B: Biomarkers: CD8+ T-cell Densities in Tumor Biopsies
Description: Fresh tumor biopsies were collected from participants in Part B of the study to assess changes in T-cell infiltration and activation within the tumor microenvironment. Tumor tissue was evaluated for CD8⁺ T-cell densities. The tumor tissue samples were collected at screening (archival metastasis and archival primary samples) and during the study (fresh samples).
Time Frame: At screening and Cycle 3 Day 1
Population: Safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Overall number analyzed = participants with data available for analysis. Number analyzed=number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells per millimetre square (cells/mm^2)
Groups:
- Part B1: Metastatic Melanoma Expansion Cohort: Participants with CPI experienced second line and beyond metastatic melanoma received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B2: NSCLC Expansion Cohort 1: Participants with CPI and platinum experienced second- or third-line PD-L1 positive NSCLC received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B4: SCLC Expansion Cohort: Participants with CPI-naïve SCLC with prior failure of, progression on, or intolerance to standard therapy received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
- Part B5: ESCC Expansion Cohort: Participants with CPI-naïve ESCC received 2100 mg, lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days)
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 25 | 19 | 5 | 7
cells per millimetre square (cells/mm^2)
  Archival Metastasis Samples: number analyzed (Participants) | 7 | 1 | 0 | 0
  Archival Metastasis Samples | 215.16 (319.52) | 29.51 (NA) — Since only 1 participant was analyzed, the SD could not be calculated. |  |
  Archival Primary Samples: number analyzed (Participants) | 2 | 5 | 0 | 3
  Archival Primary Samples | 374.92 (530.17) | 764.26 (470.25) |  | 275.02 (347.75)
  Fresh Sample 1 | 1090.51 (1001.71) | 765.44 (986.47) | 221.87 (363.76) | 510.21 (601.10)
  Fresh Sample 2: number analyzed (Participants) | 19 | 8 | 1 | 3
  Fresh Sample 2 | 912.58 (1089.90) | 790.76 (462.38) | 288.21 (NA) — Since only 1 participant was analyzed, the SD could not be calculated. | 322.23 (256.74)

10. Secondary Outcome: Parts A and B: Time to Maximum Observed Serum Concentration (Tmax) of Lomvastomig
Time Frame: Predose, half infusion, end of infusion (EOI), 0.5, 2, 4, and 8 hours postdose on Cycle 1 Day 1 and Cycle 5 Day 1, and on Cycles 1 and 5 Days 2, 3, 4, 5, 8, and 12, and predose on Day 1 of Cycles 2 and 6 (1 cycle = 14 days)
Population: Pharmacokinetic (PK) population included all participants who have received at least one dose of study treatment and who have data from at least one post-dose sample. Overall number analyzed = participants with data available for analysis. Number analyzed = participants with data available for analysis at the specified timepoint.
Measure: Median (Full Range); unit: days
Groups:
- Part A: Lomvastomig 2100 mg (Extension Cohort 1): Participants received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days). This cohort was initiated after the safety assessment of Cohort "Part A: Lomvastomig 2100 mg".
- Part A: Lomvastomig 2100 mg (Extension Cohort 2): Participants received 2100 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days). This cohort was initiated after the safety assessment of Cohort "Part A: Lomvastomig 2100 mg (Extension Cohort 1)".
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
days
  Cycle 1 | 0.09 [0.09 to 0.17] | 0.09 [0.09 to 1] | 0.125 [0.09 to 0.17] | 0.17 [0.09 to 0.26] | 0.17 [0.17 to 0.25] | 0.09 [0.09 to 0.19] | 0.175 [0.17 to 0.25] | 0.18 [0.09 to 0.28] | 0.17 [0.04 to 1.24] | 0.1 [0.04 to 0.18] | 0.17 [0.09 to 0.91] | 0.17 [0.08 to 0.25]
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 0.16 [0.16 to 0.16] | 0.17 [0.09 to 0.25] | 2.5 [1 to 4.01] | 3.57 [1.12 to 6.02] | 0.17 [0.17 to 0.17] | 0.17 [0.17 to 0.17] | 0.21 [0.09 to 0.22] | 0.215 [0.09 to 0.23] | 0.1 [0 to 0.98] | 0.1 [0.02 to 3.13] | 0.11 [0.03 to 0.11] | 0.1 [0.01 to 0.88]

11. Secondary Outcome: Parts A and B: Maximum Observed Serum Concentration (Cmax) of Lomvastomig
Time Frame: as for outcome 10
Population: PK population included all participants who have received at least one dose of study treatment and who have data from at least one post-dose sample. Overall number analyzed = participants with data available for analysis. Number analyzed = participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliters (µg/mL)
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
micrograms/milliliters (µg/mL)
  Cycle 1 | 21.5 (40.0) | 61.7 (25.2) | 148 (18.5) | 408 (5.7) | 530 (20.8) | 518 (8.8) | 575 (29.4) | 740 (14.4) | 791 (43.3) | 704 (26.2) | 726 (16.1) | 754 (24.5)
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 20.2 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 128 (8.3) | 116 (116.9) | 546 (14.8) | 781 (30.8) | 1600 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 1500 (0.0) | 1520 (17.5) | 1420 (32.6) | 1270 (33.1) | 1240 (23.0) | 1280 (25.7)

12. Secondary Outcome: Parts A and B: Maximum Observed Serum Concentration Dose Normalized (Cmax_D) of Lomvastomig
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter/milligram(µg/mL/mg)
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
microgram/milliliter/milligram(µg/mL/mg)
  Cycle 1 | 0.307 (40.0) | 0.294 (25.3) | 0.24 (18.5) | 0.34 (5.7) | 0.295 (20.9) | 0.246 (8.8) | 0.274 (29.4) | 0.352 (14.3) | 0.377 (43.2) | 0.335 (26.2) | 0.346 (16.1) | 0.359 (24.4)
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 0.777 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 0.608 (8.4) | 0.188 (117.0) | 0.455 (14.8) | 0.434 (30.8) | 0.762 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 0.714 (0.0) | 0.725 (17.5) | 0.675 (32.6) | 0.607 (33.0) | 0.592 (22.9) | 0.609 (25.8)

13. Secondary Outcome: Parts A and B: Time to Last Non-zero Concentration (Tlast) of Lomvastomig
Description: For participants who experienced an adverse event (AE) following infusion with lomvastomig, a delay of the next administration for up to two cycles was acceptable to allow for resolution of toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 2 or lower for hematological toxicities or Grade 1 or lower for non-hematological toxicities (with the exception of a toxicity considered as not related to study drug). In the case of a delayed administration, the predose PK sample for Day 1 of Cycles 2 and/or 6 could have been collected up to 28 days after the end of the previous treatment cycle.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
days
  Cycle 1 | 14 [13.9 to 14] | 14 [13.9 to 14] | 14 [13.9 to 14.1] | 14 [11.8 to 14.2] | 14 [11 to 14.1] | 14 [4.06 to 14.1] | 14.1 [13.9 to 14.2] | 14 [6.97 to 14.3] | 14 [6.07 to 16] | 14 [10.1 to 42] | 14 [13.9 to 22.1] | 14 [10.9 to 28]
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 16.9 [16.9 to 16.9] | 14 [14 to 14] | 14.1 [14 to 14.1] | 14.1 [14 to 14.1] | 15 [14.1 to 16] | 14 [14 to 14] | 14 [14 to 28] | 14.5 [13.9 to 16] | 14 [13.8 to 20.2] | 14 [13.9 to 22] | 14.5 [12.9 to 17] | 14.2 [13.9 to 21]

14. Secondary Outcome: Parts A and B: Last Non-zero Concentration (Clast) of Lomvastomig
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
µg/mL
  Cycle 1 | 5.52 (23.6) | 21.4 (9.2) | 40.4 (43.2) | 116 (17.0) | 147 (39.1) | 157 (43.2) | 157 (29.4) | 245 (29.3) | 217 (38.2) | 184 (54.1) | 194 (24.8) | 216 (46.1)
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 2.16 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 62.2 (14.5) | 59.7 (37.4) | 267 (8.8) | 415 (24.6) | 661 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 549 (22.0) | 678 (32.7) | 520 (49.6) | 495 (39.2) | 470 (59.0) | 533 (44.3)

15. Secondary Outcome: Parts A and B: Area Under the Curve From Dosing to Last Concentration (AUClast) of Lomvastomig
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*micrograms/milliliters (day*µg/mL)
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
day*micrograms/milliliters (day*µg/mL)
  Cycle 1 | 140 (37.8) | 426 (16.0) | 927 (28.8) | 2540 (22.1) | 3040 (31.6) | 2700 (52.0) | 3700 (26.8) | 4880 (30.0) | 4700 (27.9) | 4600 (27.3) | 4720 (25.7) | 5200 (24.4)
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 114 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 1200 (8.0) | 1120 (73.6) | 5470 (17.3) | 6620 (13.6) | 12200 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 13800 (28.0) | 14200 (28.4) | 11500 (43.5) | 11700 (38.1) | 9910 (39.5) | 11700 (28.7)

16. Secondary Outcome: Parts A and B: Area Under the Curve From Dosing to 336 Hours Post-dose (AUC0-336 Hrs) of Lomvastomig
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part A: Lomvastomig 2100 mg (Extension Cohort 1) | Part A: Lomvastomig 2100 mg (Extension Cohort 2) | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 4 | 4 | 11 | 38 | 25 | 15 | 16
day*µg/mL
  Cycle 1 | 140 (37.8) | 427 (15.9) | 932 (29.0) | 2600 (17.4) | 3120 (26.6) | 3180 (17.3) | 3680 (26.9) | 5060 (20.0) | 4730 (24.0) | 4550 (29.6) | 4590 (20.2) | 5150 (25.4)
  Cycle 5: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 6 | 21 | 11 | 4 | 9
  Cycle 5 | 105 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 1190 (7.7) | 1110 (74.2) | 5440 (17.6) | 6260 (21.3) | 12300 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation could not be calculated. | 11700 (1.3) | 13700 (26.4) | 11200 (41.1) | 11200 (36.1) | 9650 (41.5) | 11100 (33.6)

17. Secondary Outcome: Part A: Receptor Occupancy (RO) of Lomvastomig, Assessed Via an Ex-Vivo Assay
Description: Blood samples were collected from participants in Part A of the study and different types of immune cells were assessed by flow cytometry for the percentage of receptor occupancy (RO) by lomvastomig. RO (or drug coverage) is used to quantify the binding of the therapeutic to its target on the cell surface. The RO of lomvastomig was determined on cells that were positive (+) for CD3+, CD4+, CD56+/16+, and CD8+.
Time Frame: Predose and EOI: Day 1 of Cycles 1 and 5; Predose: Day 1 of Cycles 2, 3, and 9; Postdose: Day 8 of Cycles 1 and 5 (1 cycle is 14 days); study completion (28 days after last dose; up to 39.7 months); SFU (60 days after last dose; up to 40.8 months)
Population: Safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Overall number analyzed = participants with data available for analysis. Number analyzed = participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent occupancy
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 18
percent occupancy
  CD3+: Predose on Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 0 | 18
  CD3+: Predose on Cycle 1 Day 1 | 41.80 (37.87) | 36.23 (26.52) | 34.77 (7.79) | 0.28 (0.55) |  | 14.37 (21.43)
  CD3+: EOI on Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 4 | 3 | 18
  CD3+: EOI on Cycle 1 Day 1 | 70.43 (46.32) | 93.22 (3.03) | 106.48 (5.25) | 98.73 (12.28) | 97.47 (10.11) | 95.69 (24.36)
  CD3+: Postdose on Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 4 | 1 | 15
  CD3+: Postdose on Cycle 1 Day 8 | 108.47 (4.50) | 99.03 (14.31) | 105.33 (19.23) | 90.10 (15.62) | 91.30 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 102.53 (20.01)
  CD3+: Predose on Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 1 | 13
  CD3+: Predose on Cycle 2 Day 1 | 105.13 (9.63) | 95.53 (4.74) | 92.80 (15.65) | 93.17 (4.25) | 100.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.30 (12.10)
  CD3+: Predose on Cycle 3 Day 1: number analyzed (Participants) | 3 | 5 | 1 | 2 | 1 | 13
  CD3+: Predose on Cycle 3 Day 1 | 100.33 (8.21) | 90.62 (9.67) | 52.20 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 92.90 (11.46) | 96.90 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 105.48 (25.17)
  CD3+:Predose on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 6
  CD3+:Predose on Cycle 5 Day 1 | 62.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.20 (5.10) | 124.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated.. | 140.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 94.90 (8.77) | 92.72 (48.52)
  CD3+: EOI on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 7
  CD3+: EOI on Cycle 5 Day 1 | 82.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 95.23 (16.77) | 128.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 106.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 82.20 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 95.77 (12.49)
  CD3+: Postdose on Cycle 5 Day 8: number analyzed (Participants) | 1 | 3 | 0 | 2 | 2 | 9
  CD3+: Postdose on Cycle 5 Day 8 | 206.70 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 93.17 (12.72) |  | 96.95 (4.31) | 106.90 (12.30) | 108.28 (15.34)
  CD3+: Predose on Cycle 9 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 1 | 2 | 4
  CD3+: Predose on Cycle 9 Day 1 | 117.90 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 92.45 (6.58) |  | 101.20 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 101.40 (0.00) | 113.55 (20.00)
  CD3+: SFU: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 2
  CD3+: SFU | 98.70 (1.84) | 128.10 (18.38) |  | 95.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 90.25 (2.05) | 98.35 (2.33)
  CD3+: Study Completion: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 8
  CD3+: Study Completion | 86.35 (7.71) | 88.93 (6.90) | 94.75 (21.57) | 98.95 (9.69) | 100.50 (0.71) | 96.73 (9.11)
  CD4+: Predose on Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 15
  CD4+: Predose on Cycle 1 Day 1 | 39.93 (29.46) | 37.77 (32.40) | 30.07 (1.95) | 5.70 (7.96) |  | 16.37 (20.93)
  CD4+: EOI on Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 4 | 3 | 18
  CD4+: EOI on Cycle 1 Day 1 | 68.60 (47.94) | 92.28 (5.74) | 107.58 (3.57) | 99.80 (11.72) | 102.67 (12.71) | 96.63 (25.26)
  CD4+: Postdose on Cycle 1 Day 8: number analyzed (Participants) | 2 | 4 | 4 | 4 | 1 | 15
  CD4+: Postdose on Cycle 1 Day 8 | 97.65 (16.48) | 101.40 (16.85) | 106.53 (21.55) | 92.18 (13.53) | 88.40 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 103.77 (28.34)
  CD4+: Predose on Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 1 | 13
  CD4+: Predose on Cycle 2 Day 1 | 98.77 (16.42) | 94.28 (5.71) | 97.23 (10.71) | 91.33 (9.38) | 102.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.77 (12.11)
  CD4+: Predose on Cycle 3 Day 1: number analyzed (Participants) | 2 | 5 | 1 | 2 | 1 | 13
  CD4+: Predose on Cycle 3 Day 1 | 94.40 (3.82) | 93.38 (7.51) | 60.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 90.00 (9.48) | 100.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 98.44 (33.59)
  CD4+: Predose on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 5
  CD4+: Predose on Cycle 5 Day 1 | 68.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 96.27 (7.48) | 144.70 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 165.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 95.65 (6.15) | 112.00 (17.78)
  CD4+: EOI on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 7
  CD4+: EOI on Cycle 5 Day 1 | 103.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 91.80 (18.83) | 130.30 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 114.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 79.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 94.86 (20.02)
  CD4+: Postdose on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 0 | 2 | 2 | 8
  CD4+: Postdose on Cycle 5 Day 1 | 146.70 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 95.60 (11.36) |  | 97.60 (8.77) | 108.10 (14.42) | 102.90 (16.18)
  CD4+: Predose on Cycle 9 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 1 | 2 | 4
  CD4+: Predose on Cycle 9 Day 1 | 108.20 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 93.55 (15.06) |  | 105.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 99.15 (5.16) | 109.45 (12.18)
  CD4+: SFU: number analyzed (Participants) | 1 | 2 | 0 | 1 | 2 | 2
  CD4+: SFU | 88.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 129.45 (31.47) |  | 94.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 92.15 (2.19) | 98.30 (5.23)
  CD4+: Study Completion: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 8
  CD4+: Study Completion | 87.05 (8.70) | 95.07 (4.60) | 98.40 (24.04) | 97.65 (7.99) | 100.95 (1.34) | 97.98 (10.69)
  CD56+/16+:Predose on Cycle 1 Day 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 2 | 18
  CD56+/16+:Predose on Cycle 1 Day 1 | 57.53 (49.85) | 88.43 (37.59) | 88.87 (11.20) | 37.73 (65.36) | 73.55 (27.93) | 88.31 (43.57)
  CD56+/16+:EOI on Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 4 | 3 | 18
  CD56+/16+:EOI on Cycle 1 Day 1 | 86.80 (29.86) | 100.32 (22.37) | 107.25 (10.70) | 90.58 (73.61) | 117.73 (38.13) | 103.07 (27.26)
  CD56+/16+:Postdose on Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 3 | 2 | 17
  CD56+/16+:Postdose on Cycle 1 Day 8 | 98.43 (56.80) | 123.60 (49.67) | 90.18 (9.67) | 67.53 (17.54) | 101.90 (39.74) | 106.75 (64.75)
  CD56+/16+:Predose on Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 4 | 3 | 2 | 16
  CD56+/16+:Predose on Cycle 2 Day 1 | 100.00 (0.00) | 89.10 (3.99) | 47.83 (36.63) | 34.83 (30.25) | 112.15 (35.85) | 101.78 (20.05)
  CD56+/16+:Predose on Cycle 3 Day 1: number analyzed (Participants) | 2 | 5 | 2 | 2 | 3 | 14
  CD56+/16+:Predose on Cycle 3 Day 1 | 20.00 (28.28) | 60.76 (36.97) | 42.40 (59.96) | 55.35 (31.18) | 71.83 (18.61) | 115.75 (57.23)
  CD56+/16+:Predose on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 2 | 1 | 2 | 8
  CD56+/16+:Predose on Cycle 5 Day 1 | 100.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 82.10 (21.67) | 50.80 (5.23) | 25.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 90.35 (2.05) | 107.54 (26.49)
  CD56+/16+:EOI on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 2 | 1 | 1 | 9
  CD56+/16+:EOI on Cycle 5 Day 1 | 73.90 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 73.33 (64.07) | 32.15 (25.24) | 75.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 91.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.64 (11.65)
  CD56+/16+:Postdose on Cycle 5 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 2 | 2 | 8
  CD56+/16+:Postdose on Cycle 5 Day 8 | 3000.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 108.97 (15.53) | 0.00 (0.00) | 83.35 (23.55) | 100.50 (3.96) | 107.59 (31.13)
  CD56+/16+:Predose on Cycle 9 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 1 | 2 | 5
  CD56+/16+:Predose on Cycle 9 Day 1 | 194.10 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 25.00 (35.36) |  | 105.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 89.00 (4.67) | 98.86 (18.06)
  CD56+/16+: SFU: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  CD56+/16+: Study Completion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  CD8+: Predose on Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 15
  CD8+: Predose on Cycle 1 Day 1 | 36.37 (40.21) | 36.23 (23.99) | 53.37 (18.41) | 0.00 (0.00) |  | 17.60 (25.08)
  CD8+: EOI on Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 4 | 3 | 17
  CD8+: EOI on Cycle 1 Day 1 | 74.37 (44.30) | 95.60 (4.75) | 106.88 (11.27) | 97.18 (12.62) | 94.80 (19.83) | 99.85 (25.09)
  CD8+: Postdose on Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 4 | 1 | 15
  CD8+: Postdose on Cycle 1 Day 8 | 109.03 (9.42) | 97.48 (10.55) | 107.10 (19.15) | 91.88 (19.21) | 100.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 105.34 (23.71)
  CD8+: Predose on Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 1 | 13
  CD8+: Predose on Cycle 2 Day 1 | 113.70 (2.36) | 95.95 (3.72) | 95.13 (27.80) | 96.63 (5.83) | 95.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 98.85 (16.69)
  CD8+: Predose on Cycle 3 Day 1: number analyzed (Participants) | 3 | 5 | 1 | 2 | 1 | 12
  CD8+: Predose on Cycle 3 Day 1 | 109.13 (22.69) | 88.66 (11.84) | 58.30 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 94.50 (8.91) | 100.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 95.82 (35.78)
  CD8+: Predose on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 5
  CD8+: Predose on Cycle 5 Day 1 | 42.90 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.67 (1.15) | 110.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 115.20 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 89.15 (12.52) | 111.22 (23.82)
  CD8+: EOI on Cycle 5 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 7
  CD8+: EOI on Cycle 5 Day 1 | 75.00 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 100.17 (8.18) | 117.60 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 94.30 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 88.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 93.90 (15.31)
  CD8+: Postdose on Cycle 5 Day 8: number analyzed (Participants) | 1 | 3 | 0 | 2 | 2 | 9
  CD8+: Postdose on Cycle 5 Day 8 | 305.30 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 89.33 (10.45) |  | 92.55 (4.17) | 106.05 (10.25) | 103.67 (9.40)
  CD8+: Predose on Cycle 9 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 1 | 2 | 4
  CD8+: Predose on Cycle 9 Day 1 | 118.50 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 101.25 (1.77) |  | 94.40 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 107.90 (9.33) | 109.20 (23.66)
  CD8+: SFU: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 2
  CD8+: SFU | 108.75 (7.85) | 134.55 (0.78) |  | 93.90 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 88.75 (2.19) | 100.75 (1.06)
  CD8+: Study Completion: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 8
  CD8+: Study Completion | 86.45 (19.16) | 91.00 (23.91) | 103.00 (26.02) | 99.90 (11.88) | 101.25 (1.20) | 93.83 (10.53)

18. Secondary Outcome: Part B: Number of Participants With at Least One AE by Highest Severity, Graded According to the NCI CTCAE v5.0
Description: as for outcome 2
Time Frame: From signing of informed consent form up to 90 days after last treatment administration (up to 46.2 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
Number analyzed (Participants) | 38 | 26 | 15 | 16
Participants
  AEs (Any Grade) | 34 | 25 | 15 | 16
  Grade 1 AE | 7 | 5 | 2 | 0
  Grade 2 AE | 15 | 10 | 5 | 4
  Grade 3 AE | 11 | 9 | 8 | 10
  Grade 4 AE | 1 | 0 | 0 | 1
  Grade 5 AE | 0 | 1 | 0 | 1

19. Secondary Outcome: Part A: ORR as Determined by Investigator Using RECIST v1.1
Description: ORR was defined as the percentage of participants with an objective tumor response of CR or PR as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD.
Time Frame: Cycle 1 Day 1 then every 8 weeks for the first year; every 12 weeks thereafter until disease progression or treatment discontinuation (whichever occurs last), initiation of a new line of therapy or death (Up to 39.7 months) (Cycle length= 14 days)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19
percentage of participants | 0 (0.00) [0.00 to 63.16] | 0 (0.00) [0.00 to 45.07] | 0 (0.00) [0.00 to 52.71] | 0 (0.00) [0.00 to 52.71] | 0 (0.00) [0.00 to 52.71] | 21.1 (7.53) [7.53 to 41.91]

20. Secondary Outcome: Part A: DCR as Determined by Investigator Using RECIST v1.1
Description: DCR was defined as the percentage of participants with an objective tumor response of CR, PR or SD as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 19
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19
percentage of participants | 33.3 [1.70 to 86.46] | 40.0 [7.64 to 81.07] | 0 [0.00 to 52.71] | 50.0 [9.76 to 90.24] | 25.0 [1.27 to 75.14] | 42.1 [22.97 to 63.19]

21. Secondary Outcome: Part A: DOR as Determined by Investigator Using RECIST v1.1
Description: DOR was calculated for participants who had a best confirmed OR of CR/PR. DOR was defined as time from first occurrence of a documented OR until the time of documented PD or death from any cause, whichever occurs first as determined by investigator assessment using RECIST v1.1. CR=the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR=at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD=at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Data for participants without PD or death from any cause as of the data cut-off date were censored at the time of the last tumor assessment.
Time Frame: From first occurrence of documented OR up to disease progression or death (Up to 39.7 months) (Cycle length= 14 days)
Population: Efficacy population included participants in the safety population who received at least one dose of study drug and who had at least one baseline and one on-study tumor assessment. Overall number analyzed included participants with OR i.e., responders.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Part A: Lomvastomig 210 mg: Participants received 210 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter or until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4
months |  |  |  |  |  | 13.8 [5.6 to NA] — The upper limit of the 90% CI was not estimable due to insufficient number of participants with events.

22. Secondary Outcome: Part A: PFS as Determined by Investigator Using RECIST v1.1
Description: as for outcome 6
Time Frame: From initiation of study treatment (Cycle 1 Day 1) until disease progression or death (Up to 39.7 months) (Cycle length= 14 days)
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part A: Lomvastomig 70 mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 4 | 19
months | 1.8 [1.7 to NA] — The upper limit of the 90% CI was not estimable due to insufficient number of participants with events. | 2.0 [1.9 to 5.4] | 1.6 [1.0 to NA] — The upper limit of the 90% CI was not estimable due to insufficient number of participants with events. | NA [0.7 to NA] — The median and upper limit of the 90% CI was not estimable due to insufficient number of participants with events. | 1.8 [0.6 to NA] — The upper limit of the 90% CI was not estimable due to insufficient number of participants with events. | 1.9 [1.7 to 3.5]

ADVERSE EVENTS:
Time Frame: Part A: From signing of informed consent form up to 60 days after last treatment administration (up to 41.7 months); Part B: From signing of informed consent form up to 90 days after last treatment administration (up to 46.2 months)
Description: Safety population included all participants who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Part A: Lomvastomig 70mg: Participants received 70 mg of lomvastomig, as an IV infusion on Cycle 1 Day 1 and Q2W thereafter until disease progression, unacceptable toxicities, or withdrawal of consent, whichever occurred first (Cycle length = 14 days).
Arm/Group | Part A: Lomvastomig 70mg | Part A: Lomvastomig 210 mg | Part A: Lomvastomig 615 mg | Part A: Lomvastomig 1200 mg | Part A: Lomvastomig 1800 mg | Part A: Lomvastomig 2100 mg | Part B1: Metastatic Melanoma Expansion Cohort | Part B2: NSCLC Expansion Cohort 1 | Part B4: SCLC Expansion Cohort | Part B5: ESCC Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/5 | 4/4 | 2/4 | 2/4 | 13/19 | 26/38 | 18/26 | 13/15 | 8/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5 | 1/4 | 1/4 | 1/4 | 7/19 | 6/38 | 8/26 | 4/15 | 10/16
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 4/4 | 4/4 | 3/4 | 17/19 | 34/38 | 24/26 | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lomvastomig 70mg (N=3) | Part A: Lomvastomig 210 mg (N=5) | Part A: Lomvastomig 615 mg (N=4) | Part A: Lomvastomig 1200 mg (N=4) | Part A: Lomvastomig 1800 mg (N=4) | Part A: Lomvastomig 2100 mg (N=19) | Part B1: Metastatic Melanoma Expansion Cohort (N=38) | Part B2: NSCLC Expansion Cohort 1 (N=26) | Part B4: SCLC Expansion Cohort (N=15) | Part B5: ESCC Expansion Cohort (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gallbladder abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
False positive investigation result (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lomvastomig 70mg (N=3) | Part A: Lomvastomig 210 mg (N=5) | Part A: Lomvastomig 615 mg (N=4) | Part A: Lomvastomig 1200 mg (N=4) | Part A: Lomvastomig 1800 mg (N=4) | Part A: Lomvastomig 2100 mg (N=19) | Part B1: Metastatic Melanoma Expansion Cohort (N=38) | Part B2: NSCLC Expansion Cohort 1 (N=26) | Part B4: SCLC Expansion Cohort (N=15) | Part B5: ESCC Expansion Cohort (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 6 (10) | 5 (7) | 6 (7) | 5 (6) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Thyroid disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 5 (7) | 2 (2) | 4 (4) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 7 (8) | 6 (6) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (9) | 6 (6) | 1 (1) | 2 (2) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (4)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (4) | 8 (10) | 3 (6) | 2 (2) | 5 (5)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 9 (15) | 3 (3) | 1 (1) | 2 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (7) | 16 (20) | 8 (8) | 5 (5) | 1 (2)
Chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 6 (8) | 5 (6) | 4 (4) | 7 (8)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 4 (7) | 6 (6) | 0 (0) | 2 (2)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Accidental underdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Human chorionic gonadotropin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 9 (10) | 4 (4) | 4 (4) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 7 (8) | 0 (0) | 1 (1) | 2 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 4 (4) | 4 (4) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 3 (4)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 5 (5) | 2 (2) | 3 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 7 (7) | 4 (6) | 6 (6) | 2 (2) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 1 (1) | 4 (4) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 3 (3) | 0 (0) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03708328/Prot_SAP_000.pdf